CLINICAL TRIAL: NCT00634530
Title: Impact of a Nutritional Intervention Program for Weight Control During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Márcia Regina Vitolo, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: vitolo4
Record Dates: First submitted 2008-03-10; First posted 2008-03-13 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Pregnancy Complications; Weight Gain
Keywords: Pregnancy; Prenatal Care; Weight; Nutritional Status
MeSH Terms: conditions — Pregnancy Complications; Weight Gain; Body Weight | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- I, Intervention (Other)
  Interventions: Behavioral: Dietary Advice

INTERVENTIONS:
Behavioral: Dietary Advice — The specific dietary advices according to nutritional status. Main advices: reduction of fat and sugar intake, increase of total energy, dairy intake of vegetables and fruits.

SUMMARY:
This is a randomized clinical trial for evaluate the impact of a nutritional intervention in the weight control of pregnant women according to the nutritional status, and consequently, the reduction of pregnancy complications.

The sample of this study will be composed by 318 pregnant women in the pre-natal care unit of the Health Center in Viamão city / Rio Grande do Sul, including women between the 10th and 25th weeks of gestation, aged up to 35 years old. The eligible pregnant women will be invited by the fieldworks to participated in the trial after be informed about the overall aims of the study. These women willing to participate will be randomly allocated to either the intervention or control group. The intervention group received specific guidelines about feeding practices appropriate to each nutritional status.

Data on pregnant women will be collected through a questionnaire in both groups, and to assess the food intake, three 24-hour food recall will be applied in the interventional group and two recall in the control group, in initial and final gestational period. In all appointments pregnant women of the two groups will be weight and classified according to Body Mass Index of pre-gestational (BMI).

The dietary advices will be elaborated by the author of the project and nutrition graduation students of Federal University of Health Science of Porto Alegre.

ELIGIBILITY:
Inclusion Criteria:

* Women between the 10th and 25th weeks of gestation
* To concern in the prenatal care group in basic health unit

Exclusion Criteria:

* Pregnant with diseases that require specific treatment at the onset enrollment (HIV, diabetes, hypertension and anemia)
* Women 36 years or older.

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 318 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Adequated weight gain during pregnancy. | one year

SECONDARY OUTCOMES:
Prematurity, low birth weight and pregnancy complications. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Márcia R Vitolo, Doctor, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Health Center, Viamão, Rio Grande do Sul, Brazil